CLINICAL TRIAL: NCT01994824
Title: Preemptive Therapy of Graft-vs-Host Disease Using Rabbit Antithymocyte Globulin
Brief Title: Preemptive Therapy of GVHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trend was observed toward higher mortality among the patients receiving the intervention Thymoglobulin on day 8 after hematopoietic cell transplantation.
Sponsor: University of Calgary (Other)
Collaborators: University of Alberta (Other); Alberta Health services (Other)
Responsible Party: Principal Investigator, Jan Storek, Professor of Medicine, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PreemptiveATG
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Graft-vs-host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention arm (Experimental): Transplant recipients will have IL15 and IL2Ra measured on day 7. If at risk for significant GVHD, the patient will get rabbit antithymocyte globulin, 3 mg/kg on day 8.
  Patients from this intervention/experimental arm will be compared to historical and concurrent controls (no ATG on day 8).
  Interventions: Drug: rabbit antithymocyte globulin

INTERVENTIONS:
Drug: rabbit antithymocyte globulin — Thymoglobulin, 3 mg/kg, will be given on day 8 posttransplant to patients at high risk of significant GVHD per day 7 IL15 and IL2Ra levels.
  Other Names: Thymoglobulin

SUMMARY:
Graft-vs-host disease (GVHD) causes substantial mortality, morbidity and poor quality of life after blood or marrow transplantation (BMT). In Alberta, we use antithymocyte globulin (ATG, given on days -2, -1 and 0) in addition to methotrexate and cyclosporine for GVHD prophylaxis. In spite of that, ~40% patients develop significant GVHD (grade 2-4 acute GVHD or chronic GVHD needing systemic immunosuppressive therapy). ATG at the dose we typically use (4.5 mg/kg) is relatively non-toxic. At higher doses, ATG could increase the likelihood of posttransplant infections or relapse. Thus an extra dose of ATG (on top of the routine 4.5 mg/kg) might be justified only for patients at high risk of developing significant GVHD. In our experience, low serum level of interleukin-15 (IL15) and high serum level of interleukin-2 receptor alpha (IL2Ra) on day 7 predict development of significant GVHD. Here we will test whether, compared to historical/concurrent controls, an extra dose of ATG (3 mg/kg on day 8) given to patients with low IL15 or high IL2Ra on day 7 reduces the incidence of significant GVHD, and improves survival free of relapse and GVHD, and quality of life.

DETAILED DESCRIPTION:
Blood for IL15 and IL2Ra determination will be drawn in the morning of day 7 (10 ml red top tube). IL15 and IL2Ra levels will be measured in Storek/Khan Lab by enzyme-linked immunosorbent assay (ELISA) as described (Pratt LM et al: BMT 2013). Storek/Khan Lab staff will report the IL15 and IL2Ra levels to the Bone Marrow Transplant ward (Unit 57, Foothills Medical Centre) no later than in the morning of day 8. If the IL15 level is <31 ng/L or the IL2Ra level is >4500 ng/L, the physician caring for the patient on the ward will order Thymoglobulin, 3 mg/kg intravenously, to be infused over 4-8 hours on day 8. The dose is based on actual body weight, and is rounded to the nearest vial (Thymoglobulin is supplied in 25 mg vials) except if the rounding would result in >5% difference from the calculated dose. Unit 57 standard practice will be followed for the infusion of ATG (see Standard Operation Procedure BMTS40153 ["ATG Administration"]). Premedication for ATG will include methylprednisolone 40 mg IVPB, acetaminophen 1000 mg PO and diphenhydramine 50 mg IVPB. Acetaminophen 1000 mg PO and diphenhydramine 50 mg IVPB can be repeated in 4-6 hours PRN flu-like symptoms/fever/chills. Meperidine 25-50 mg IVPB every 4 hours will be given PRN for rigors.

EVALUATIONS For the endpoint of the incidence of significant GVHD, patients will be followed per standard practice of the Alberta Blood and Marrow Transplant Program for the development of acute and chronic GVHD (www.albertahealthservices.ca/hp/if-hp-cancer-guide-bmt-manual.pdf). Per this standard practice, acute GVHD is graded according to Consensus criteria (Przepiorka D: BMT 1995) and chronic GVHD is diagnosed and graded according to NIH criteria (Filipovich AH: BBMT 2005). Significant GVHD is defined as grade 2-4 acute GVHD or chronic GVHD needing systemic immunosuppressive therapy.

For the endpoint of survival free of significant GVHD and relapse, relapse will be defined by standard criteria (eg, >5% marrow blasts by morphology in case of acute leukemia).

For the endpoint of quality of life at 2 years (21-27 months) posttransplant, Short Form 36 will be used.

ELIGIBILITY:
Inclusion Criteria:

1. First allogeneic hematopoietic cell transplantation (second transplants are rare, typically performed for relapse of leukemia, in which case the likelihood of relapse is high, and there is the theoretical risk of increasing the likelihood further with ATG).
2. Conditioning including ATG 4.5 mg/kg (the predictive value of IL15 and IL2Ra levels was determined in patients whose conditioning included 4.5 mg/kg or ATG).
3. Age >17 (the predictive value of IL15 and IL2Ra levels has not been studied in children).

Exclusion Criteria:

1. Nonmyeloablative conditioning (possible risk of ATG increasing relapse).
2. Active viral infection (risk of worsening of the viral infection with ATG).
3. Neutropenic fever with hypotension. In such case, the ATG can be given on day 9 (instead of day 8) if patient no longer has hypotension.
4. Hypoxemia. In such case, the ATG can be given on day 9 (instead of day 8) if patient no longer has hypoxemia.
5. History of anaphylactic reaction to Thymoglobulin or another rabbit blood protein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of significant GVHD | 2 years

SECONDARY OUTCOMES:
Survival free of relapse and significant GVHD | 2 years
Quality of life measured by SF36 | 2 years
  Short Form 36

CONTACTS AND LOCATIONS:
Overall Officials: Jan Storek, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Health Services-CancerControl / University of Calgary / University of Alberta (Edmonton), Calgary, Alberta, Canada

REFERENCES:
- [Derived] Khanolkar RA, Kalra A, Kinzel M, Pratt LM, Dharmani-Khan P, Chaudhry A, Williamson TS, Daly A, Morris DG, Khan FM, Storek J. A biomarker-guided, prospective, phase 2 trial of pre-emptive graft-versus-host disease therapy using anti-thymocyte globulin. Cytotherapy. 2021 Nov;23(11):1007-1016. doi: 10.1016/j.jcyt.2021.06.003. Epub 2021 Aug 6. PMID 34373186